CLINICAL TRIAL: NCT04863339
Title: Tranexamic Acid for Blood Loss Minimization in Endoscopic Pituitary Surgery: A Double-Blind Randomized Controlled Trial
Brief Title: Tranexamic Acid for Blood Loss Minimization in Endoscopic Pituitary Surgery
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Challenges in recruitment
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 20-2267
Record Dates: First submitted 2021-04-23; First posted 2021-04-28 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Pituitary Tumor; Blood Loss; Surgery
MeSH Terms: conditions — Pituitary Neoplasms; Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: Participants randomized to receive the investigational product vs placebo during a single study encounter.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The only staff with access to randomization codes will be our study statistician who created the randomization table and our investigational drug services pharmacy who is preparing the investigational product.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tranexamic Acid (Experimental): Participants in the Tranexamic Acid arm will receive a dose of Tranexamic Acid.
  Interventions: Drug: Tranexamic acid
- Placebo (Placebo Comparator): Patients in the placebo arm will receive a saline placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tranexamic acid — Single preoperative dose of 1 gram of Tranexamic Acid in 100 mL of saline given 0-30 minutes prior to surgery.
  Arms: Tranexamic Acid
Drug: Placebo — Single preoperative dose of 100 mL of saline placebo given 0-30 minutes prior to surgery.
  Arms: Placebo

SUMMARY:
This trial is to determine the effect of Tranexamic Acid (TXA) on blood loss during endoscopic pituitary surgery. The hypothesis of this study is that TXA will reduce blood loss during surgery compared to a placebo. To answer this hypothesis, the investigators are conducting a randomized controlled trial in which half of participants will receive TXA and half will receive placebo (saline) in a double blind fashion.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing endoscopic pituitary surgery at UNC

Exclusion Criteria:

* Clival invasion
* Giant pituitary tumor (>4 cm)
* Revision pituitary surgery
* Prior sinus surgery
* Lund McKay score > 3
* Active thromboembolic disease
* Coagulopathy
* Concomitant pro-thrombotic medications
* Concomitant use of anti-coagulants or anti-platelet agents
* Subarachnoid hemorrhage
* History of severe hypersensitivity to Tranexamic Acid

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-03 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Mean Blood Loss | Time between incision and surgical closure, an average of 3 to 3.5 hours
  Blood loss measured in mL

SECONDARY OUTCOMES:
Intra-operative Surgical Visibility - Wormald Scale Score | Duration of operation, up to 4 hours
  Wormald scale (0-10):
  The Wormald grading scale is a validated grading tool to measure visual field quality during endoscopic endonasal procedures.
  Lower scores indicate less bleeding and better surgical visibility.
  0 = No bleeding (optimal)
  1. = 1-2 points of blood ooze
  2. = 3-4 points of ooze
  3. = 5-6 points of ooze
  4. = 7-8 points of ooze
  5. = 9-10 points of ooze
  6. = >10 points of ooze, obscuring field
  7. = Mild field bleeding with slow post-nasal accumulation
  8. = Moderate field bleeding with moderate post-nasal accumulation
  9. = Moderate-severe field bleeding with rapid post-nasal accumulation
  10. = Severe bleeding (worst) with nose filling rapidly
  These measurements will take place 6 times. During hours 1, 2, 3, and 4 of the surgery, as well as during sphenoidotomy and durotomy.

OTHER OUTCOMES:
Incidence of Venous Thromboembolism | from time of intervention administration through 1 week after surgery
  Absolute number of incident venous thromboembolism
Mean Duration of Surgery | Time between incision and surgical closure, an average of 3 to 3.5 hours
  Measured in hours

CONTACTS AND LOCATIONS:
Overall Officials: Brent Senior, MD, Principal Investigator — UNC Chapel Hill

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 12 to 24 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol
Time Frame: 12 to 24 months following publication
Access Criteria: Requests for IPD can be made by email and will be reviewed by the PI. The study protocol and deidentified data can be provided for scientific analyses performed by physicians and researchers affiliated with academic institutions.

REFERENCES:
- [Background] Roberts I, Shakur H, Coats T, Hunt B, Balogun E, Barnetson L, Cook L, Kawahara T, Perel P, Prieto-Merino D, Ramos M, Cairns J, Guerriero C. The CRASH-2 trial: a randomised controlled trial and economic evaluation of the effects of tranexamic acid on death, vascular occlusive events and transfusion requirement in bleeding trauma patients. Health Technol Assess. 2013 Mar;17(10):1-79. doi: 10.3310/hta17100. PMID 23477634
- [Background] Ping WD, Zhao QM, Sun HF, Lu HS, Li F. Role of tranexamic acid in nasal surgery: A systemic review and meta-analysis of randomized control trial. Medicine (Baltimore). 2019 Apr;98(16):e15202. doi: 10.1097/MD.0000000000015202. PMID 31008946
- [Background] Heyns M, Knight P, Steve AK, Yeung JK. A Single Preoperative Dose of Tranexamic Acid Reduces Perioperative Blood Loss: A Meta-analysis. Ann Surg. 2021 Jan 1;273(1):75-81. doi: 10.1097/SLA.0000000000003793. PMID 32224739
- [Background] Jahanshahi J, Hashemian F, Pazira S, Bakhshaei MH, Farahani F, Abasi R, Poorolajal J. Effect of topical tranexamic acid on bleeding and quality of surgical field during functional endoscopic sinus surgery in patients with chronic rhinosinusitis: a triple blind randomized clinical trial. PLoS One. 2014 Aug 18;9(8):e104477. doi: 10.1371/journal.pone.0104477. eCollection 2014. PMID 25133491
- [Background] Mebel D, Akagami R, Flexman AM. Use of Tranexamic Acid Is Associated with Reduced Blood Product Transfusion in Complex Skull Base Neurosurgical Procedures: A Retrospective Cohort Study. Anesth Analg. 2016 Feb;122(2):503-8. doi: 10.1213/ANE.0000000000001065. PMID 26554461